CLINICAL TRIAL: NCT01296087
Title: A Phase II Multicenter, Randomized, Double-Blind,Parallel Group, Placebo-Controlled Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetic Parameters of TC-6987 in Subjects With Persistent Mild to Moderate Asthma
Brief Title: TC-6987 for the Treatment of Mild to Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TC-6987-23-CRD-001
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
Keywords: Asthma; Mild to Moderate Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-6987 (Experimental)
  Interventions: Drug: TC-6987
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-6987 — TC-6987 50 mg capsule given once daily on Days 1 to 28
  Arms: TC-6987
Drug: Placebo — Matching placebo capsule given once daily on Days 1 to 28
  Arms: Placebo

SUMMARY:
This study is designed to determine whether TC-6987 improves respiratory function in subjects with asthma by reducing airway hyper-responsiveness and inflammation.

DETAILED DESCRIPTION:
Asthma is a common, chronic inflammatory disorder of the airways that affects an estimated 20 to 22 million people in the United States. It is characterized by variable and recurring symptoms, notably airflow obstruction, bronchial hyperresponsiveness, and an underlying inflammation. The bronchospasm is caused by inflammation of the muscles surrounding the air passageways, making them smaller, thus more difficult for air to freely move in and out of the lungs. Cardinal symptoms of asthma include coughing, chest tightness, shortness of breath and wheezing. These symptoms are often more severe in the morning and late night, and usually reversible with medications. Clinically, asthma is typically classified according to the frequency of symptoms, forced expiratory volume in 1 second (FEV1), and peak expiratory flow rate.

The rationale for this Phase II proof of concept study is to demonstrate that TC-6987 improves respiratory function in subjects with asthma, compared to placebo, as measured by the Baseline FEV1 on Day 1 compared to the End-of-Treatment FEV1 on Day 28 or Early Withdrawal (EW); and also to assess the safety and tolerability profile of TC-6987 in subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of persistent mild to moderate asthma requiring at least 3 months of daily treatment with inhaled corticosteroids (ICS).
2. A FEV1 value at Screening that is 60-90% of predicted FEV1.
3. Age 18 to 65, males or females.

Exclusion Criteria:

1. Diagnosis or presence of other pulmonary diseases including chronic obstructive pulmonary disease (COPD) and emphysema.
2. Previous life-threatening asthma, such as asthma requiring intubation or ICU admission for asthma.
3. Prolonged hospitalization for asthma within the past year (emergency room treatments using nebulized beta-agonists is permitted).
4. Not able and willing to stop the use of long-acting beta-agonists (LABAs), cromolyn sodium, methylxanthines, anticholinergic agents, leukotriene inhibitors, or any other non-ICS or non-SABA prescription or over-the-counter anti-asthma medication, including antihistamines, during Screening and during the Study.
5. Use of moderate to strong cytochrome P450 3A4 (CYP3A4) inhibitors.
6. Use of oral steroids within the last 1 month, or use of >/= 3 steroid bursts in the last 12 months.
7. History of upper respiratory tract infection (URI) requiring treatment during the last month prior to Screening.
8. Tobacco use within 3 months prior to Screening, or > 5 pack-year lifetime tobacco use.
9. Use of smoking cessation therapy within 3 months prior to Screening.
10. Uncontrolled Gastroesophageal reflux disease (GERD). Subjects on a stable dose of non-prescription or prescription medications who have been symptom free for 4 wks prior to screening are eligible.
11. History within past 6 months of alcohol abuse or illicit drug abuse.
12. Myocardial infarction within 12 months prior to Screening.
13. Known hypothyroidism, vitamin B12, or folic acid deficiency.
14. Known systemic infection (HBV, HCV, HIV, TB).
15. FSH level of < 35 IU/L and a LH level < 25 IU/L.
16. Urine cotinine level > 50 ng/ml.
17. Body Mass Index (BMI) <15 and >35.
18. Participation in another clinical trial in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 status on Day 28 compared to baseline as a function of treatment (TC-6987 versus placebo) | Day 28
  Co-primary efficacy endpoints:
  1. the change in FEV1 from pre dose on Day 1 to pre dose on Day 28
  2. the change in FEV1 from pre dose on Day 1 to 2 h post dose on Day 28

SECONDARY OUTCOMES:
Number of Asthma Control Days | Day 1
  Number of Asthma Control Days from 14 days prior to Day 1, compared to the 14 days prior to Day 28, as a function of Treatment
Decrease in FEV1 after methacholine dose as a function of treatment | Day 29
  Percentage of patients in which methacholine dose decreases FEV1 by 20% (PC20) at Day 29 compared to Day -1
Number of Asthma Control Days | Day 28
  Number of Asthma Control Days from 14 days prior to Day 1, compared to the 14 days prior to Day 28, as a function of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Winder, MD, Principal Investigator — Toledo Center for Clinical Research
Locations (21):
- United States (21):
  - Clinical research Center of Alabama, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - California Allergy and Asthma Medical Group, Inc., Los Angeles, California
  - California Allergy & Asthma Medical Group, Palmdale, California
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - Avail Clinical Research LLC, DeLand, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Florida Pulmonary Research Institute, Inc., Winter Park, Florida
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy & Asthma Clinical Research Center, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Altoona Lung Specialists, Altoona, Pennsylvania
  - Allergy & Asthma Research of New Jersey, Inc., Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Pioneer Research Solutions, Houston, Texas
  - Paragon Research, San Antonio, Texas
  - Utah Clinical Trials, LLC, Salt Lake City, Utah
  - VA Adult & Pediatric Allergy & Asthma PC, Richmond, Virginia
  - Pulmornary Consultants, PLLC, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin